CLINICAL TRIAL: NCT05235048
Title: Single Tooth Extraction in Damaged Alveoli and Implant Site Development Randomized Controlled Clinical Trial Comparing Socket Preservation and Reconstruction Surgery to Spontaneous Healing
Brief Title: Single Tooth Extraction in Damaged Alveoli and Implant Site Development:TootToo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The European Research Group on Periodontology (ERGOPerio) (Network)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERGOPerio 15-01
Record Dates: First submitted 2020-01-11; First posted 2022-02-10 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Tooth Extraction Status Nos
Keywords: Alveolar ridge preservation; Tooth extraction; Dental implant
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Intervention Model Description: This will be a parallel group, standard of care-controlled, assessor-blind, randomized, multicenter, superiority clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Independent outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of care control (Placebo Comparator): Tooth extraction and spontaneous healing
  Interventions: Procedure: Tooth extraction
- Socket seal with CT graft (Experimental): Tooth extraction and socket sealing with autologous connective tissue graft
  Interventions: Procedure: Tooth extraction; Procedure: Tooth extraction and socket seal with connective tissue graft
- Socket seal with CT graft and bone replacement graft (Experimental): Tooth extraction and socket sealing with autologous connective tissue graft and positioning of bone replacement graft in coronal portion of the socket
  Interventions: Procedure: Tooth extraction; Procedure: Tooth extraction and socket seal with connective tissue graft; Procedure: Tooth extraction and socket seal with BRG and connective tissue graft and
- Tooth extraction and socket sealing and BRG with membrane (Experimental): Tooth extraction and socket sealing with autologous connective tissue graft and positioning of bone replacement graft in coronal portion of the socket and positioning of collagen membrane
  Interventions: Procedure: Tooth extraction; Procedure: Tooth extraction and socket seal with connective tissue graft; Procedure: Tooth extraction and socket seal with BRG and connective tissue graft and; Procedure: Tooth extraction and socket seal with membrane placement, BRG and connective tissue graft

INTERVENTIONS:
Procedure: Tooth extraction — Atraumatic tooth extraction without flap elevation
Procedure: Tooth extraction and socket seal with connective tissue graft — Atraumatic tooth extraction without flap elevation and seal of the alveolar socket with connective tissue graft (microsurgery)
  Arms: Socket seal with CT graft; Socket seal with CT graft and bone replacement graft; Tooth extraction and socket sealing and BRG with membrane
Procedure: Tooth extraction and socket seal with BRG and connective tissue graft and — Atraumatic tooth extraction without flap elevation, position of a bone replacement graft into the socket and seal of the alveolar socket with connective tissue graft (microsurgery)
  Arms: Socket seal with CT graft and bone replacement graft; Tooth extraction and socket sealing and BRG with membrane
Procedure: Tooth extraction and socket seal with membrane placement, BRG and connective tissue graft — Atraumatic tooth extraction without flap elevation, position of a collagen membrane and bone replacement graft into the socket and seal of the alveolar socket with connective tissue graft (microsurgery)
  Arms: Tooth extraction and socket sealing and BRG with membrane

SUMMARY:
It is unclear what is the best approach to implant site development after tooth extraction when the pathology leading to extraction has damaged the alveolus. The main objective of this study is to assess if socket preservation and/or reconstruction surgery provides a clinical benefit in terms of ability to place an implant in a prosthetically guided position in such clinical conditions.

The PICO question therefore is:

In patients requiring single tooth extraction what is the benefit of socket preservation/reconstruction surgery with respect to spontaneous healing in terms of feasibility and ease of implant surgery?

DETAILED DESCRIPTION:
This will be a parallel group, standard of care-controlled, assessor-blind, randomized, multicenter, clinical trial.

The statistical design will be a superiority trial in terms of the primary outcome with reference to the standard of care control (spontaneous healing).

Primary outcome:

Possibility to place an implant in a prosthetically driven position with or without bone or soft tissue augmentation 16-20 weeks after tooth extraction, evaluated at planning with cone beam CT and confirmed at surgery.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy. No contraindications to elective oral surgery
* All pathologies requiring single tooth extraction with adjacent teeth (or implant) with the presence of at least one third of the alveolus.
* Evidence of subject ability to achieve good oral hygiene and control gingivitis in the whole of the dentition (FMPS<25% and FMBS<25%)
* Ability to understand study procedures and to comply with them for the entire length of the study. Ability and willingness to give informed consent.

Exclusion Criteria:

* Presence of frank purulence or acute abscess at the time of extraction
* Presence of bone resorption of one or more walls of the alveolus extending to the apical third of the socket
* Self reported current smoking exceeding 20 cigarettes/day or pipe or cigar smoking
* Presence of medical contraindications to elective surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Possibility to place dental implant | 16-20 weeks
  The possibility to place a dental implant in a prosthetically driven position (with or without bone or soft tissue augmentation) 16-20 weeks after tooth extraction will be evaluated with a dedicated planning software using cone beam CT data and and digital scanning according to standard clinical practice
Surgeon's confirmation of the ability to place a dental implant | 16-20 weeks
  Confirmation during the surgery of the ability to actually insert the implant in a prosthetically driven position with or without the need for soft or hard-tissue augmentation.

SECONDARY OUTCOMES:
Vertical change in bone height at the deepest point in the socket | 16-20 weeks
  Bone fill of the socket evaluated at the time of dental implant placement as change in the distance between a customized surgical stent and the bottom of the alveolus using a periodontal probe (difference between baseline and 16-20 week healing)
Vertical change in bone height at the buccal bone crest | 16-20 weeks
  Bone fill of the socket evaluated at the time of dental implant placement as change in the distance between a customized surgical stent and the bottom of the alveolus using a periodontal probe (difference between baseline and 16-20 week healing)
Vertical change in bone height at the crest of adjacent teeth | 16-20 weeks
  Harm to bone of adjacent teeth measured by clinical attachment level loss and trans gingival probing.
Radiographic bone changes | 16-20 weeks
  Bone fill of the socket measured on routine intraoral radiographs
Change in keratinized tissue width between baseline and insertion of prosthetic crown | 16-20 weeks
  Soft tissue preservation assessed as millimetre of keratinised tissue as measured with a periodontal probe
Need for additional bone augmentation at the time of implant placement (and/or implant uncovering, if submerged healing) | 16-20 weeks
  Need for additional augmentation assessed by the surgeon during implant placement
Wound healing index | 1-4 weeks
  Early healing assessed with standardized composite healing index by dentist
OHIP-14 | 1-2 weeks
  Oral health related quality of life standard instrument (questionnaire) - 5 point Likert scale with greater scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Cortellini, MD, Study Director — Investigator

IPD SHARING:
Plan to Share IPD: No
Data will not be shared